CLINICAL TRIAL: NCT05322213
Title: The Effects of THC on Glucose Metabolism and Endothelial Function in Subjects With Type 2 Diabetes
Brief Title: THC Effects on Glucose in Type 2 Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Center for Medicinal Cannabis Research (Other)
Responsible Party: Principal Investigator, Jeremy Pettus, MD, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 802153
Record Dates: First submitted 2022-03-30; First posted 2022-04-11 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: THC
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Intervention Model Description: Single-Center, double-blind, placebo-controlled, crossover study.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active THC (Active Comparator): Daily, inhaled, flexible dose of cannabis product with THC.
  Interventions: Drug: THC; Drug: Placebo
- Placebo Cannabis (Placebo Comparator): Daily, inhaled, flexible dose of cannabis product without THC.
  Interventions: Drug: THC; Drug: Placebo

INTERVENTIONS:
Drug: THC — 2-Week, once daily, flexible dose, inhaled THC
  Other Names: Cannabis
Drug: Placebo — 2-Week, once daily, flexible dose, inhaled placebo

SUMMARY:
This study will examine the effects THC has on Glucose Metabolism and Endothelial Functioning in participants with Type 2 Diabetes. The participants will complete blood tests and tests to measure energy expenditure, CVD risks, and glucose metabolism. These tests will be performed prior to start of treatment and again after 2-weeks of treatment with the THC or placebo.

DETAILED DESCRIPTION:
A single-center, double-blind, placebo-controlled, cross-over study designed to evaluate the effects of THC on glucose metabolism and endothelial functioning in individuals with type 2 diabetes. To accomplish the specific AIMS proposed, a single clinical trial will be conducted in which a maximum of 30 subjects with T2D, who are otherwise healthy, will be treated with THC and matching placebo in a cross-over study design. Each treatment period will be 2 weeks in duration with metabolic and endothelial assessments done post-therapy. Subjects will be randomized on a 1:1 basis to either receive either THC or placebo for the first 2 weeks of therapy. Then following a 4-week washout, they will receive the opposite investigational product for the second 2 weeks of therapy. Subjects will remain on their standard treatment for T2D throughout the entire course of the study. There will be a total of 10 study visits and subjects will be enrolled for approximately 16 weeks.

1. Screening - Complete consenting process, complete medical history and physical exam, review of current medications, collect height/weight, vital signs, ECG and fasting laboratory (blood and urine) tests.
2. Visit 2 - Treatment Session 1 Start - Collect weight, vital signs and fasting laboratory tests. Receive investigational product and training on its use.
3. Visit 3 - Monitory investigational product compliance and adjust dosing.
4. Visit 4 - Complete endothelial function tests including flow mediated dilation and EndoPat, complete vital signs, weight and laboratory tests for safety.
5. Visit 5 - Complete a 2-Step Hyperinsulinemic/Euglycemic clamp and Indirect Calorimetry. Begin 4-week washout.
6. Visit 6 - Treatment Session 2 Start - Collect weight, vital signs and receive investigational product and training on its use.
7. Visit 7 - Monitory investigational product compliance and adjust dosing.
8. Visit 8 - Complete endothelial function tests including flow mediated dilation and EndoPat, complete vital signs, weight and laboratory tests for safety.
9. Visit 9 - Complete a 2-Step Hyperinsulinemic/Euglycemic clamp and Indirect Calorimetry. Discontinue use of investigational product.
10. Safety Follow-up - Collect weight, vital signs, ECG and fasting laboratory tests. Receive investigational product and training on its use.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 21-70 years old at the time of screening.
* Females of non-child bearing potential must be ≥ 1 year post-menopausal or documented as being surgically sterile. Females of child bearing potential must agree to use two methods of contraception during the entire study.
* Male subjects must be willing to use clinically acceptable method of contraception during the entire study.
* Have a clinical diagnosis of Type 2 Diabetes on a stable medication regimen for at least 3 months.
* BMI > 25 kg/m2).
* HbA1c < 10%).
* Negative urine toxicology result at screening visit.
* Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

* History or presence of any clinically significant illness, as detected by history, physical examination, and/or laboratory tests, that might put the participant at increased risk of adverse events (e.g., history of psychotic disorder, clinically significant mood and/or anxiety disorder, liver, or renal disease).
* No prior history of myocardial infarction, stroke or heart failure.
* Whole blood donation of 1 pint (500 mL) within 8 weeks prior to Screening. Donations of plasma, packed RBCs, platelets or quantities less than 500 mL are allowed at investigator discretion.
* Hemoglobin < 9g/dL.
* Liver enzymes ≥ 2 times upper normal limit and/or clinical signs/symptoms consistent with liver disease, including but not limited to nausea, vomiting, jaundice, itching, abdominal pain, or edema.
* History of clinically significant adverse events associated with cannabis intoxication (e.g., severe anxiety and panic, paranoia and psychosis, sustained tachycardia, or severe hypotension).
* History of seizures, head trauma, or other history of CNS insult that could predispose the participant to seizures.
* Use of any THC containing products within 30 days prior to the screening visit.
* Current use of tobacco products.
* Individuals who are pregnant or lactating/breastfeeding.
* Current use of insulin to treat Type 2 Diabetes.
* Unable or unwilling to follow the study protocol or who are non-compliant with screening appointments or study visits.
* Any other condition(s) that might reduce the chance of obtaining study data, or that might cause safety concerns, or that might compromise the ability to give truly informed consent.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in Glucose Uptake | 6 weeks
  The change in glucose uptake from placebo treatment to THC treatment as measure by the hyperinsulinemic/euglycemic clamp.
Change in Vascular Endothelial Function | 6 weeks
  The change in vascular endothelial function from placebo treatment to THC treatment as measured by flow mediated dilation (brachial artery diameter).
Change in Vascular Endothelial Function | 6 weeks
  The change in vascular endothelial function from placebo treatment to THC treatment as measured by reactive hyperemia-peripheral arterial tonometry (reactive hyperemia index).

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Altman Clinical & Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No